CLINICAL TRIAL: NCT07056101
Title: Evaluation of Pain Perception Using Computer-Controlled Local Anaesthesia Delivery With Different Injection Speeds Versus Conventional Anaesthesia for Maxillary Primary Molars: A Randomized Controlled Trial
Brief Title: "Study of Pain Perception Using Computer-Controlled Versus Conventional Local Anaesthesia in Children Undergoing Molar Extraction
Acronym: CCLAD-Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarek MHD kher al saka amini (Other)
Responsible Party: Sponsor-Investigator, Tarek MHD kher al saka amini, DOCTOR, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GENI-CCLAD VS CA
Record Dates: First submitted 2025-06-19; First posted 2025-07-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dental Phobia; Dental Anxiety; Dental Anesthesia; Dental Anesthesia Efficacy
Keywords: GENI Device; Pain Perception; Local Anesthesia Technique; Articaine; Computer-Controlled Local Anesthesia; Dental Injections

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1:1:1 ratio to one of four parallel groups: three receiving local anesthesia using the GENI computer-controlled device at different injection speeds (high, moderate, or low), and one receiving anesthesia via conventional syringe. Each participant will receive only one intervention throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GENI High-Speed Injection (Experimental): Participants in this arm will receive local anesthesia using the GENI computer-controlled local anesthesia delivery (CCLAD) device set to high-speed injection mode. Buccal and intrapapillary infiltration will be administered using 4% articaine with 1:100,000 epinephrine. The injection will be performed by the principal investigator following a standardized technique. Pain perception will be evaluated immediately after injection.
  Interventions: Device: GENI High-Speed Injection
- GENI Moderate-Speed Injection (Experimental): Participants in this arm will receive local anesthesia using the GENI computer-controlled local anesthesia delivery (CCLAD) device set to moderate-speed injection mode. The injection will include buccal and intrapapillary infiltration using 4% articaine with 1:100,000 epinephrine. The procedure will be performed by the principal investigator using a standardized technique. Pain perception will be assessed immediately following the injection.
  Interventions: Device: GENI Moderate-Speed Injection
- GENI Low-Speed Injection (Experimental): Participants in this arm will receive local anesthesia using the GENI computer-controlled local anesthesia delivery (CCLAD) device set to low-speed injection mode. Buccal and intrapapillary infiltration will be administered using 4% articaine with 1:100,000 epinephrine. The injection will be performed by the principal investigator following a standardized protocol. Pain perception will be evaluated using subjective, objective, and physiological measures.
  Interventions: Device: GENI Low-Speed Injection
- A Conventional dental Syringe (Active Comparator): Participants in this arm will receive local anesthesia using a traditional metal aspirating dental syringe (C-K JECT) with a short 30-gauge needle. Buccal and intrapapillary infiltration will be performed using 4% articaine with 1:100,000 epinephrine, following a standardized injection technique. The procedure will be conducted by the principal investigator. Pain perception will be assessed immediately after the injection using subjective, objective, and physiological parameters.
  Interventions: Device: A conventional dental syringe

INTERVENTIONS:
Device: A conventional dental syringe — The conventional dental syringe (C-K JECT) is a manual, metal aspirating syringe commonly used for local anesthesia administration in dental procedures. In this study, the device is used to perform buccal and intrapapillary infiltration using 4% articaine with 1:100,000 epinephrine. Injections are delivered manually at a standardized rate by the principal investigator. This arm serves as the active comparator to evaluate differences in pain perception between traditional syringe injections and those delivered via a computer-controlled device.
  Arms: A Conventional dental Syringe
Device: GENI High-Speed Injection — The GENI device is a computer-controlled local anesthesia delivery system that automates the injection process using pressure feedback to regulate flow. In this arm, the device is set to high-speed mode to deliver the anesthetic solution at the fastest available flow rate. Buccal and intrapapillary infiltration is performed using 4% articaine with 1:100,000 epinephrine. The procedure is carried out by the principal investigator using a standardized technique. Pain perception is assessed following injection to evaluate the impact of delivery speed on patient experience.
  Arms: GENI High-Speed Injection
Device: GENI Moderate-Speed Injection — The GENI device is a computer-controlled local anesthesia delivery system designed to regulate flow and pressure during injection using real-time feedback. In this arm, the device is set to moderate-speed mode, delivering anesthetic at an intermediate flow rate. Buccal and intrapapillary infiltration is performed using 4% articaine with 1:100,000 epinephrine. The injection is administered by the principal investigator using a standardized technique. This group is used to assess the impact of moderate-speed delivery on pain perception and physiological response in pediatric patients.
  Arms: GENI Moderate-Speed Injection
Device: GENI Low-Speed Injection — The GENI device is a computer-controlled local anesthesia delivery system that maintains precise control over injection pressure and flow. In this arm, the device is set to low-speed mode, delivering the anesthetic solution at the slowest available rate to minimize tissue pressure and potential discomfort. Buccal and intrapapillary infiltration is administered using 4% articaine with 1:100,000 epinephrine. The injection is performed by the principal investigator using a standardized technique. This group evaluates whether low-speed delivery reduces pain perception and improves patient comfort compared to faster injection speeds and conventional methods.
  Arms: GENI Low-Speed Injection

SUMMARY:
This clinical trial aims to compare pain perception in children during dental procedures when using a computer-controlled local anesthesia device versus a traditional syringe. Children aged 6 to 8 years who need maxillary primary molar extraction will be randomly assigned to one of four groups: three groups using different speeds of the GENI computer-controlled device, and one group using a conventional syringe. The study will assess pain using facial expression scales and physiological measures such as heart rate. The goal is to find a more comfortable method for delivering anesthesia to pediatric dental patients.

DETAILED DESCRIPTION:
This is a parallel-design randomized controlled clinical trial evaluating pain perception during local anesthesia administration in children undergoing extraction of maxillary primary molars. The study compares the use of a computer-controlled local anesthesia delivery system (GENI) at three different injection speeds-high, moderate, and low-with conventional syringe-based anesthesia.

Children aged 6 to 8 years who meet the inclusion criteria will be randomly allocated to one of four groups using a computer-generated randomization sequence. Standardized injection techniques will be applied in all groups. The primary outcome is subjective pain, assessed using the Wong-Baker FACES Pain Rating Scale. Secondary outcomes include objective behavioral pain assessments using the FLACC scale and physiological responses such as heart rate and oxygen saturation measured with a pulse oximeter.

All procedures will be performed by a single trained operator. The assistant supervisor will monitor randomization and data collection. Although blinding of the operator and participants is not feasible due to the nature of the devices, outcome assessors and the statistician will remain blinded to group assignment to reduce bias.

The study aims to identify whether the GENI device provides improved comfort, reduced pain, and greater cooperation among pediatric patients compared to traditional local anesthesia techniques. The results are expected to guide the development of better pain management strategies in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 6 to 8 years old
* Both sexes
* Healthy children classified as ASA I
* Children with maxillary primary molars indicated for extraction
* No previous dental experience
* Mentally capable of communication and following instructions
* No acute dental pain

Exclusion Criteria:

* Uncooperative children or those with a behavioral management problem (Frankl rating 1 or 2)
* Children with known allergies to the local anesthetic or dental materials used in the study
* Children taking medications (e.g., antibiotics, analgesics) in the previous 48 hours that may alter pain perception
* Children whose parents or legal guardians refuse to sign the informed consent form
* Children experiencing acute dental pain

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Subjective Pain Perception During Local Anesthesia Injection | Immediately after local anesthesia injection
  Pain perception will be measured using the Wong-Baker FACES Pain Rating Scale, which ranges from 0 (no pain) to 10 (worst pain). Each child will select the face that best represents their level of pain immediately following the injection. This scale is a validated tool for assessing subjective pain in pediatric patients.

SECONDARY OUTCOMES:
Objective Pain Perception During local anathesia Injection (FLACC Scale) | During local anesthesia injection(Day 1)
  Objective pain will be assessed using the FLACC Scale during the local anathesia injection . An external evaluator will observe and score facial expression,leg movement,activity,crying,and consolability.
  Unit of measure :
  Score (0-10)
Heart rate Response to Local Anesthesia injection | Baseline (within 10 minutes before injection )and during injection (Day 1)
  Heart rate will be measured using a fingertip pulse oximeter to evaluate physiological stress response. Reading will be taken before injection (baseline) and during the injection.
  Unit of measure :
  Beats per minute (bpm)
Oxygen Saturation During Local Anesthesia injection | Baseline (within 10 minutes before injection ) and during injection (Day 1)
  Oxygen saturation (%) will be measured using a fingertip pulse oximeter at baseline and during the injection to assess any change in oxygen levels as a physiological response to stress or pain.
  Unit of measure :
  Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mariam mohsen Associate Professor of Pediatric Dentistry and Dental Public, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) that underlie the results reported in the final publication (text, tables, figures, and appendices) will be made available upon reasonable request. Access will be granted to researchers with a methodologically sound proposal for secondary analysis. Data will be available beginning 6 months after publication and ending 2 years after publication.

REFERENCES:
- See also: Official website of the Faculty of Dentistry at Cairo University, providing information about academic programs, research activities, and departmental contacts related to dental studies. — https://dentistry.cu.edu.eg